CLINICAL TRIAL: NCT01806402
Title: Evaluation of the Precision and Accuracy of OCT Measurements in Retinal and Glaucoma Patients
Brief Title: Evaluation of OCT Measurements
Status: Completed | Type: Observational
Sponsor: Optovue (Industry)
Responsible Party: Sponsor
Other Study IDs: 20130104
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Assess Eye Measurements in Patients Having Retina Pathology or Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retina: Having clinical diagnosis of retina pathology
- Glaucoma: Having clinical diagnosis of glaucoma

SUMMARY:
The purpose of the study is to repeatability, reproducibility and agreement of eye measurements in retina and glaucoma patients.

DETAILED DESCRIPTION:
The purpose of the study is to repeatability, reproducibility and agreement of eye measurements in retina and glaucoma patients using OCT technology. There will be a series of measurements acquired from one eye on at least 2 different OCT devices. All testing will be completed in one visit.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criterea:

* At least 18 years of age
* Able and willing to provide consent
* Willing to complete the required examinations and visits
* Best corrected visual acuity equal or better than 20/100
* Retina subject must have clinical diagnosis of retinal pathology
* Glaucoma subjects must have clinical diagnosis of glaucoma

Exclusion Criteria:

* Unable to complete the required examinations and visits
* Poor OCT image quality as a result of media opacity, extreme refractive error or pathologies in the anterior segment
* Confounding pathology requiring surgical treatment or medical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will have retina pathology or glaucoma.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2013-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Retina thickness | Day 1

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Pacific Eye Specialists, Daly City, California
  - North Bay Eye Associates, Petaluma, California
  - West Coast Retinal Medical Group, Walnut Creek, California